CLINICAL TRIAL: NCT03172832
Title: A Multicenter Randomized Trial of Percutaneous Transhepatic Biliary Drainage vs. Endoscopic Retrograde Cholangiography for Decompression of Suspected Malignant Biliary Hilar Obstruction - the INTERCPT Trial
Brief Title: A Trial of Percutaneous vs. Endoscopic Drainage of Suspected Klatskin Tumors
Acronym: INTERCPT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual; recommended by DSMB.
Sponsor: Medical University of South Carolina (Other)
Collaborators: Yale University (Other); Virginia Commonwealth University (Other); Vanderbilt University (Other); Stony Brook University (Other); University of Southern California (Other); Case Western Reserve University (Other); Medical College of Wisconsin (Other); Dartmouth University (Other); University of Florida (Other); Northwestern University (Other); Johns Hopkins University (Other); Washington University School of Medicine (Other); University of Michigan (Other); Boston University (Other); Ohio State University (Other); Borland-Groover Clinic (Other); Methodist Health System (Other); St. Louis University (Other); Fox Chase Cancer Center (Other); Emory University (Other); Cedars-Sinai Medical Center (Other); Johns Hopkins Community Physicians (Other); University of Virginia (Other)
Responsible Party: Principal Investigator, Badih Elmunzer, Professor of Medicine, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00063825
Record Dates: First submitted 2017-05-26; First posted 2017-06-01 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Cholangiocarcinoma; Hilar Lymphadenopathy; Biliary Stricture
MeSH Terms: conditions — Cholangiocarcinoma | interventions — perfluoro-2,2,2',2'-tetramethyl-4,4'-bis(1,3-dioxolane)

STUDY DESIGN:
Intervention Model Description: Randomized comparative effectiveness trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous Transhepatic Drainage (Active Comparator): Subjects randomized to this arm will undergo PTBD as the first drainage intervention.
  Interventions: Procedure: PTBD
- Endoscopic Retrograde Cholangiography (Active Comparator): Subjects randomized to this arm will undergo ERC as the first drainage intervention.
  Interventions: Procedure: ERC

INTERVENTIONS:
Procedure: PTBD — Percutaneous access and tube placement into the bile duct
  Arms: Percutaneous Transhepatic Drainage
Procedure: ERC — Endoscopic access and stent placement in the bile duct
  Arms: Endoscopic Retrograde Cholangiography

SUMMARY:
The optimal approach to the drainage of malignant obstruction at the biliary hilum remains uncertain. This is a randomized comparative effectiveness study of percutaneous transhepatic biliary drainage (PTBD) vs. endoscopic retrograde cholangiography (ERC) as the first intervention in patients with cholestasis due to suspected malignant hilar obstruction.

DETAILED DESCRIPTION:
Both percutaneous transhepatic biliary drainage (PTBD) and endoscopic retrograde cholangiography (ERC) are accepted approaches in the management of patients with malignant obstruction at the biliary hilum. In routine clinical practice, ERC is generally favored on the basis of: 1) high technical and clinical success rates for other (non-hilar) indications; 2) the perceived safety of ERC relative to PTBD; 3) the perceived ability to perform more comprehensive tissue sampling at the time of ERC compared to PTBD; 4) the avoidance of external tubes which are often needed for PTBD; and 5) because patients with suspected malignant hilar obstruction (MHO) typically present to and are managed by gastroenterologists. However: 1) observational data suggest that PTBD is superior for achieving complete drainage of MHO1 and some guidelines recommend the percutaneous approach over ERC for Bismuth type 3 & 4 hilar strictures; 2) the generally quoted risks of PTBD are based on outdated studies and may be exaggerated; and 3) endoscopic diagnosis of indeterminate biliary strictures remains suboptimal despite the use of cholangioscopy and multi-modal sampling.

Although many patients who undergo initial ERC require subsequent PTBD for adequate drainage, no randomized trials comparing the two modalities for suspected MHO have been published. The main hypothesis is that even though PTBD will be more effective than ERC for decompression of suspected MHO, this advantage will be offset by the favorable safety profile and superior diagnostic capability of ERC. If, however, PTBD is found to be substantially superior (by a pre-specified margin) in terms of drainage, or if the potential advantages of ERC are not realized, then the existing clinical approach to MHO must be reappraised. Moreover, identifying patient and stricture characteristics that predict response to PTBD or ERC may be important for informing clinical decision-making and guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥40 (to reduce the likelihood of enrolling patients with obstruction due to primary sclerosing cholangitis)
2. Cholestatic liver function tests, including serum alkaline phosphatase level ≥ 300 IU/L and bilirubin level ≥ 3.7 mg/dL
3. Radiographic evidence of a biliary hilar stricture OR intrahepatic but no extrahepatic biliary ductal dilation

Exclusion Criteria:

1. Known radiographic evidence of a Bismuth-Corlette type 1 biliary stricture
2. Known diagnosis of primary sclerosing cholangitis without suspicion of dominant hilar stricture
3. Recent gallbladder/biliary surgery within 12 months
4. Known Mirizzi syndrome
5. Known IgG4-mediated cholangiopathy
6. Significant liver metastatic disease interfering with safe/effective PTBD
7. Significant ascites interfering with safe/effective PTBD
8. Known regional malignant-appearing adenopathy or extra-biliary mass, indicating the need for concurrent EUS-FNA
9. Prior ERCP or PTBD for hilar obstruction
10. Surgically altered luminal anatomy other than prior Billroth reconstruction or Whipple resection
11. Standard general contraindications to ERCP or PTBD (e.g. hemodynamic instability, uncorrected coagulopathy, etc.)
12. Inability or unwillingness to follow study protocol

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-08-20 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

PRIMARY OUTCOMES:
Successful biliary drainage | 2 weeks
  50% reduction in bilirubin level within 2 weeks of the study intervention without additional ERC or PTBD

SECONDARY OUTCOMES:
Alternate definition of successful biliary drainage | 6 months
  improvement in the serum bilirubin level to ≤2.5 mg/dL as a result of the index (randomization) intervention without the need for additional procedures.
Adverse events | 6 months
  Adverse events related to PTBD and ERC, defined according to standard consensus guideline documents published in the interventional radiology and gastroenterology literature respectively.
Adequate tissue diagnosis | 6 months
  A definitive diagnosis of malignancy documented in the subject's medical record.
Quality of life measure | 2-3 months after initial procedure
  Promis Global Health Scale
Quality of life measure | 2-3 months after initial procedure
  SF12 health survey

CONTACTS AND LOCATIONS:
Overall Officials: B. Joseph Elmunzer, Principal Investigator — Medical University of South Carolina
Locations (25):
- United States (25):
  - University of Southern California, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - University of Florida - Jacksonville, Jacksonville, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Boston University, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Saint Louis University, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Dartmouth University, Lebanon, New Hampshire
  - Stony Brook University, Stony Brook, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Methodist Hospital Dallas, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Kawas F, Aslanian H, Baillie J, Banovac F, Buscaglia JM, Buxbaum J, Chak A, Chong B, Cote GA, Draganov PV, Dua K, Durkalski V, Elmunzer BJ, Foster LD, Gardner TB, Geller BS, Jamidar P, Jamil LH, Keswani RN, Khashab MA, Lang GD, Law R, Lichtenstein D, Lo SK, McCarthy S, Melo S, Mullady D, Nieto J, Bayne Selby J, Singh VK, Spitzer RL, Strife B, Tarnaksy P, Taylor JR, Tokar J, Wang AY, Williams A, Willingham F, Yachimski P; In alphabetical order for the INTERCPT Study Group and the United States Cooperative for Outcomes Research in Endoscopy (USCORE). Percutaneous transhepatic vs. endoscopic retrograde biliary drainage for suspected malignant hilar obstruction: study protocol for a randomized controlled trial. Trials. 2018 Feb 14;19(1):108. doi: 10.1186/s13063-018-2473-2. PMID 29444707